CLINICAL TRIAL: NCT04274166
Title: The Efficacy and Safety of Secukinumab for the Inflammatory Phase of Pyoderma Gangrenosum
Brief Title: Secukinumab for the Inflammatory Phase of Pyoderma Gangrenosum
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Contracting never completed, closed the IRB
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00063109; Huang_IIT_CAIN457AUS24T (Other Grant/Funding Number: Novartis)
Record Dates: First submitted 2020-02-12; First posted 2020-02-18 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Pyoderma Gangrenosum
MeSH Terms: conditions — Pyoderma Gangrenosum | interventions — secukinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): 2 s.c. secukinumab 150 mg injections
  Interventions: Drug: secukinumab 150 mg (2 injections per dose

INTERVENTIONS:
Drug: secukinumab 150 mg (2 injections per dose — secukinumab 150 mg (2 injections per dose
  Other Names: secukinumab

SUMMARY:
The purpose of this research study is to find out what effects (good and bad) secukinumab has on the subject and their pyoderma gangrenosum.

Secukinumab is a type of medicine called human monoclonal antibodies. Monoclonal antibodies are proteins that recognize and attach to other specific proteins (in this case, immune system hormones called "cytokines") that your body produces. The cytokine (a "messenger" protein in the body) that secukinumab binds to and reduces the activity of is a naturally occurring cytokine called interleukin-17A (IL-17A). IL-17A is believed to be partly responsible for inflammation (pain, swelling, redness), and researchers believe that IL-17A may cause symptoms PG.

DETAILED DESCRIPTION:
This is a prospective, single center, Phase IIa study of secukinumab in the treatment of subjects diagnosed with PG. Subjects will be evaluated at Screening, Baseline (week 0), Week 1, Week 2, Week 3, Week 4, and then every 4 weeks for 24 weeks. The total duration of treatment is up to 20 weeks. Subjects may be treated for shorter durations if the lesions clear prior to week 20. Subjects will have a follow-up visit at 24 weeks, or 4 weeks after the last dose of study drug. Subjects will also have standard of care wound dressings done at each visit. Subjects will be given 300 mg of secukinumab SQ at week 0, 1, 2, 3, and 4, followed by injections every 4 weeks, for up to 20 weeks. Subjects may receive a dose increase at week 16 (if there is not at least a 25% reduction in target lesion size) to 300 mg every 2 weeks.

* Complete Blood Count (CBC), Comprehensive Metabolic panel (CMP), C- reactive protein (CRP), Erythrocyte sedimentation rate (ESR), Hepatitis panel, HIV test, Pregnancy test, and QuantiFERON gold TB test will be performed at screening. (Appendix 6)
* CBC, CMP, CRP, ESR will be performed at week 8 and week 20.
* Pain rating by Likert scale (A 10-point scale to rate the level of pain - Appendix 2), an Investigator Global Assessment (IGA) (Appendix 3), Subject Global Assessment (SGA) (Appendix 3), and Ulcer Lesion Assessment (Appendix 5) will be done at Screening, Baseline, and at Weeks 2, 4, 8, 12, 16, 20, and 24.
* Lesion photography will be done at Screening and all visits.
* Infection and adverse event assessments and concomitant medication assessments will be performed at each visit.
* Quality of life will be measured with the Dermatology Life Quality Index (DLQI) at Baseline and Week 20 (Appendix 4).

ELIGIBILITY:
Inclusion Criteria:

1. Must give written informed consent. 2. Has a diagnosis of pyoderma gangrenosum, as determined by the investigator based on the following diagnostic criteria4:

a. Diagnosis requires both major criteria and at least two minor criteria i. Major criteria

1. Rapid progression of a painful, necrolytic cutaneous ulcer with an irregular, violaceous, and undermined border
2. Other causes of cutaneous ulceration have been excluded ii. Minor criteria

1. History suggestive of pathergy or clinical finding of cribriform scarring 2. Systemic diseases associated with PG 3. Histopathologic findings (sterile dermal neutrophilia, ± mixed inflammation, ± lymphocytic vasculitis) 4. Treatment response (rapid response to systemic steroid treatment)

3. PG global assessment of moderate to severe, with at least one ulcer measuring at least 3 cm in diameter.

4. 18 years of age or greater. 5. Must require systemic therapy for their pyoderma gangrenosum, as determined by the investigator prior to Baseline. Currently prescribed low-dose corticosteroids (≤ 10 mg/day), and other medications within one week prior to investigational drug administration, may be continued with no change in dose or frequency during the study.

Exclusion Criteria:

1. Female subjects who are not postmenopausal for at least 1 year, surgically sterile, or willing to practice effective contraception during the study. Nursing mothers, pregnant women and women planning to become pregnant while on study are to be excluded.
2. Current enrollment in any investigational study in which the subject is receiving any type of drug, biologic, or non-drug therapy (participation in registry-type studies is allowed).
3. Serious local infection (e.g., cellulitis, abscess) or systemic infection (e.g., pneumonia, septicemia) within the 3 months prior to the first dose of investigational drug.
4. Treatment with another investigational drug or approved therapy for investigational use within 28 days prior to investigational drug administration.
5. Treatment with high dose (>10 mg/day) systemic steroids (prednisone) within one week prior to investigational drug administration. Treatment with cyclosporine, thalidomide, methotrexate, mycophenolate mofetil, azathioprine, or other systemic immunosuppressant agents within the 14 days prior to investigational drug administration (requirement of a 2-week washout).
6. Known HIV+, known viral hepatitis infection, known tuberculosis infection.
7. Any subject with a current or history of a malignancy in the last five years (excluding treated basal cell carcinoma).
8. Clinically significant abnormal laboratory measures at screening.
9. Known Irritable Bowel Disease-associated PG

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-05 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Efficacy - Investigator Global Assessment (IGA) | Screening visit
  Investigator Global Assessment (IGA) as measured by a 7 point scale anchored by 'Completely Clear" and "Worse"
Efficacy - Investigator Global Assessment (IGA) | Change from Screening visit to Baseline visit.
  Investigator Global Assessment (IGA) as measured by a 7 point scale anchored by 'Completely Clear" and "Worse"
Efficacy - Investigator Global Assessment (IGA) | Change from Baseline visit to Week 2.
  Investigator Global Assessment (IGA) as measured by a 7 point scale anchored by 'Completely Clear" and "Worse"
Efficacy - Investigator Global Assessment (IGA) | Change from week 2 to week 4.
  Investigator Global Assessment (IGA) as measured by a 7 point scale anchored by 'Completely Clear" and "Worse"
Efficacy - Investigator Global Assessment (IGA) | Change from Week 4 to week 8.
  Investigator Global Assessment (IGA) as measured by a 7 point scale anchored by 'Completely Clear" and "Worse"
Efficacy - Investigator Global Assessment (IGA) | Change from Week 8 to week 12.
  Investigator Global Assessment (IGA) as measured by a 7 point scale anchored by 'Completely Clear" and "Worse"
Efficacy - Investigator Global Assessment (IGA) | Change from Week 12 to week 16.
  Investigator Global Assessment (IGA) as measured by a 7 point scale anchored by 'Completely Clear" and "Worse"
Efficacy - Investigator Global Assessment (IGA) | Change from Week 16 to week 20.
  Investigator Global Assessment (IGA) as measured by a 7 point scale anchored by 'Completely Clear" and "Worse"
Efficacy - Investigator Global Assessment (IGA) | Change from Week 20 to week 24.
  Investigator Global Assessment (IGA) as measured by a 7 point scale anchored by 'Completely Clear" and "Worse"
Efficacy - Subject Global Assessment (SGA) | Baseline.
  Subject Global Assessment (SGA) as measured by a 7 point scale anchored by 'Completely Clear" and "Worse"
Efficacy - Subject Global Assessment (SGA) | Change from Baseline to week 2.
  Subject Global Assessment (SGA) as measured by a 7 point scale anchored by 'Completely Clear" and "Worse"
Efficacy - Subject Global Assessment (SGA) | Change from Week 2 to Week 4.
  Subject Global Assessment (SGA) as measured by a 7 point scale anchored by 'Completely Clear" and "Worse"
Efficacy - Subject Global Assessment (SGA) | Change from Week 4 to Week 8. .
  Subject Global Assessment (SGA) as measured by a 7 point scale anchored by 'Completely Clear" and "Worse"
Efficacy - Subject Global Assessment (SGA) | Change from Week 8 to Week 12.
  Subject Global Assessment (SGA) as measured by a 7 point scale anchored by 'Completely Clear" and "Worse"
Efficacy - Subject Global Assessment (SGA) | Change from Week 12 to Week 16.
  Subject Global Assessment (SGA) as measured by a 7 point scale anchored by 'Completely Clear" and "Worse"
Efficacy - Subject Global Assessment (SGA) | Change from Week 16 to Week 20.
  Subject Global Assessment (SGA) as measured by a 7 point scale anchored by 'Completely Clear" and "Worse"
Efficacy - Subject Global Assessment (SGA) | Change from Week 20 to Week 24.
  Subject Global Assessment (SGA) as measured by a 7 point scale anchored by 'Completely Clear" and "Worse"
Efficacy - Ulcer Lesion Assessment PG Target Lesion | Change from Screening visit, Baseline, and at Weeks 2, 4, 8, 12, 16, 20, and 24.
  Number of subjects achieving 50% improvement in PG lesion size
Efficacy - Ulcer Lesion Assessment PG Target Lesion | Change from Screening visit, Baseline, and at Weeks 2, 4, 8, 12, 16, 20, and 24.
  Number of subjects achieving resolution of inflammation with an erythema score of 0 and a border elevation of 0 on five point scales of none to very severe

CONTACTS AND LOCATIONS:
Overall Officials: William W Huang, MD. MPH, Principal Investigator — Wake Forest University Health Sciences

IPD SHARING:
Plan to Share IPD: No